CLINICAL TRIAL: NCT03487419
Title: Relationship Between Echocardiographic Left Atrial Function Assessment and Atrial Fibrillation Post-Coronary Artery Bypass Surgery
Brief Title: Echocardiographic Left Atrial Function Assessment and Atrial Fibrillation Post-Coronary Artery Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Institute, Egypt (Other Government)
Responsible Party: Principal Investigator, hossam ahmed hamed hussein, Principal Investigator, National Heart Institute, Egypt
Other Study IDs: left atrial speckle tracking
Record Dates: First submitted 2018-03-27; First posted 2018-04-04 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Atrium; Fibrillation
Keywords: left atrial echocardiography; new onset atrial fibrillation; coronary artery bypass grafting; speckle tracking echocardiography
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients develop atrial fibrillation: patients post coronary artery bypass grafting who develop atrial fibrillation post operative
- patients who not develop atrial fibrillation: patients post coronary artery bypass grafting who don't develop atrial fibrillation post operative

SUMMARY:
The aim of this study to investigate the correlation between preoperative LA function using 2D echocardiography and left atrium 2D speckle tracking strain echocardiography and the development of Post Operative AF after CABG.

the investigators chose electrocardiography as a reference standard for detection of Post Operative AF. LA dysfunction is diagnosed with Echocardiography

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common postoperative complications following cardiac surgery. This in turn translates into longer hospitalization, increased cost of hospitalization as well as association with thromboembolic events and mortality .

Despite new-onset postoperative atrial fibrillation (NoPOAF) occurring in 20-40% of patients following coronary artery bypass graft (CABG) surgery, the underlying mechanisms are not well established. However, it has been traditionally thought to be transient and benign to the patient.

Recent evidence suggests that POAF may be more 'malignant' than previously thought, associated with follow-up mortality and morbidity.

Previously, increased left atrial (LA) size and LA dysfunction have been shown to be related to the subsequent development of atrial fibrillation (AF), stroke, myocardial infarction, and heart failure.

Also, recent studies suggest that LA dysfunction caused by the effects of oxidative stress, inflammation, and atrial fibrosis, has a role. In other words, by acute functional depression, preoperative LA dysfunction may be the starting point of the development of POAF after coronary artery bypass grafting (CABG).(8) Therefore, as the improvement in the evaluation of LA function, preoperative LA dysfunction may emerge as an important component in the identification of patients with the risk of POAF after CABG surgery.

Echocardiography is the most common diagnostic method for assessing atrial function but the technique has some limitations. Traditionally, assessment of left atrial function has been performed by measuring volumes with 2D echocardiography. Additionally, it can be assessed with transmitral Doppler and pulmonary vein Doppler. Recently, an alternative method has been incorporated, namely, measurement of myocardial deformation with color tissue Doppler-derived strain.

However, this method has several limitations, such as suboptimal reproducibility, angle-dependence, signal artifacts and the fact that it only measures regional strain and does not obtain information about the curved portion of the atrial roof. To overcome these limitations in the quantification of atrial function, the use of speckle tracking echocardiography (STE) strain has been proposed. This technique is not derived from Doppler but rather from 2D echocardiography, it is angle-independent, and allows us to measure global as well as regional atrial strain. STE is a new technique of 2D echocardiography image analysis that allows the study of regional atrial myocardial deformation expressed by a dimensionless parameter.

2-dimensional (2D) speckle tracking strain imaging is a feasible and reproducible technique for the assessment of LA function by evaluating LA deformation dynamics.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with preoperative sinus rhythm who were referred for elective isolated CABG (no other concomitant cardiac or extracardiac procedures).

  * Patient age more than18 years old.

Exclusion Criteria:

* • Any type of arrhythmia other than sinus.

  * Hyperthyroidism or hypothyroidism.
  * Renal failure requiring hemodialysis .
  * Moderate to severe valvular heart disease.
  * Current use of antiarrhythmic drugs .
  * Recent myocardial infarction within a month before surgery.
  * Patient with redo CABG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adult patients with preoperative sinus rhythm who were referred for elective isolated CABG (no other concomitant cardiac or extracardiac procedures) were enrolled. Standard transthoracic echocardiography and left atrial 2D speckle tracking strain echocardiography were performed preoperatively. After surgery, patients received continuous electrocardiography (ECG) monitoring throughout hospitalization in the coronary care unit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Development of new onset atrial fibrillation post coronary artery bypass grafting surgery during ICU stay and hospital stay till discharge and its relation to left atrial function assessed by echocardiography | baseline
  assessment of left atrium function by echocardiography and its relation to incidence of new onset atrial fibrillation during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Institute, Cairo, Kit Kat, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Echahidi N, Pibarot P, O'Hara G, Mathieu P. Mechanisms, prevention, and treatment of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Feb 26;51(8):793-801. doi: 10.1016/j.jacc.2007.10.043. PMID 18294562
- [Result] Haghjoo M. Pharmacological and nonpharmacological prevention of atrial fibrillation after coronary artery bypass surgery. J Tehran Heart Cent. 2012 Winter;7(1):2-9. Epub 2012 Feb 28. PMID 23074627
- [Result] Levy D, Kannel WB. Postoperative atrial fibrillation and mortality: do the risks merit changes in clinical practice? J Am Coll Cardiol. 2004 Mar 3;43(5):749-51. doi: 10.1016/j.jacc.2003.12.011. No abstract available. PMID 14998611
- [Result] Borde D, Gandhe U, Hargave N, Pandey K, Mathew M, Joshi S. Prediction of postoperative atrial fibrillation after coronary artery bypass grafting surgery: is CHA 2 DS 2 -VASc score useful? Ann Card Anaesth. 2014 Jul-Sep;17(3):182-7. doi: 10.4103/0971-9784.135841. PMID 24994728
- [Result] Mariscalco G, Engstrom KG. Postoperative atrial fibrillation is associated with late mortality after coronary surgery, but not after valvular surgery. Ann Thorac Surg. 2009 Dec;88(6):1871-6. doi: 10.1016/j.athoracsur.2009.07.074. PMID 19932252
- [Result] Abhayaratna WP, Seward JB, Appleton CP, Douglas PS, Oh JK, Tajik AJ, Tsang TS. Left atrial size: physiologic determinants and clinical applications. J Am Coll Cardiol. 2006 Jun 20;47(12):2357-63. doi: 10.1016/j.jacc.2006.02.048. PMID 16781359
- [Result] Elahi MM, Flatman S, Matata BM. Tracing the origins of postoperative atrial fibrillation: the concept of oxidative stress-mediated myocardial injury phenomenon. Eur J Cardiovasc Prev Rehabil. 2008 Dec;15(6):735-41. doi: 10.1097/HJR.0b013e328317f38a. PMID 19020458
- [Result] Her AY, Kim JY, Kim YH, Choi EY, Min PK, Yoon YW, Lee BK, Hong BK, Rim SJ, Kwon HM. Left atrial strain assessed by speckle tracking imaging is related to new-onset atrial fibrillation after coronary artery bypass grafting. Can J Cardiol. 2013 Mar;29(3):377-83. doi: 10.1016/j.cjca.2012.06.006. Epub 2012 Aug 15. PMID 22902158
- [Result] Cianciulli TF, Saccheri MC, Lax JA, Bermann AM, Ferreiro DE. Two-dimensional speckle tracking echocardiography for the assessment of atrial function. World J Cardiol. 2010 Jul 26;2(7):163-70. doi: 10.4330/wjc.v2.i7.163. PMID 21160748
- [Result] Vianna-Pinton R, Moreno CA, Baxter CM, Lee KS, Tsang TS, Appleton CP. Two-dimensional speckle-tracking echocardiography of the left atrium: feasibility and regional contraction and relaxation differences in normal subjects. J Am Soc Echocardiogr. 2009 Mar;22(3):299-305. doi: 10.1016/j.echo.2008.12.017. PMID 19258177